CLINICAL TRIAL: NCT00323635
Title: A Parallel, Double-blind Comparison of Tolterodine vs. Placebo Treatments for Nocturia in Postmenopausal Women.
Brief Title: A Comparison of Tolterodine and Placebo Treatments on Nocturnal Frequency and Sleep Quality in Women After Menopause.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: New department chairman instructed PI to discontinue study.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Quentin Rodney Regestein, MD, Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-P-000960
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Urinary Incontinence
Keywords: nocturia; urinary incontinence; overactive bladder; tolterodine; sleep; sleep disorder; menopause; midlife women; psychological tests
MeSH Terms: conditions — Urinary Incontinence; Nocturia; Urinary Bladder, Overactive; Sleep Wake Disorders | interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolterodine (Experimental): Tolterodine 4 mg q.d. X 8 weeks
  Interventions: Drug: tolterodine
- Placebo (Placebo Comparator): A capsule of identical to tolterodine in taste, smell and appearance that contains no tolterodine
  Interventions: Drug: tolterodine

INTERVENTIONS:
Drug: tolterodine — tablet, 4 mg, daily, 1 month
  Other Names: Detrol

SUMMARY:
This study is being done to compare frequency of urination during the night when women take tolterodine tablets vs. when they take placebo tablets.

We will also measure whether between these two treatment conditions there are any differences in women's sleep, mood and performance on cognitive tests.

DETAILED DESCRIPTION:
From midlife onwards, about half of women complain of poor sleep quality. One possible reason might be an increased frequency of need to urinate during the night. Women feel more frequent urges to urinate when structures that support the bladder become more lax. Tolterodine is a drug that can raise the threshold for volume of urine that accumulates in the bladder before the urge to urinate arises.

Many factors determine how people say they sleep, such as their sleep as recorded by sleep-measuring instruments, how closely they notice their night's sleep, whether they are generally prone to make positive or negative judgments or to have a lot or a few body symptoms.

In this study, women between ages 45 to 65 who are past the menopause and who are frequently bothered by the need to urinate during the night will take either tolterodine or placebo tablets for 8 weeks. During the last week they will record the hours they slept and the quality of their sleep each morning. They will wear a device on their wrist through the week that continuously records whether they are asleep or awake. During three nights of the week they will record the volume of urine whenever they urinate. At the end of the week they will complete questionnaires about their mood and take some computerized tests that measure their alertness. Thereafter they will repeat these procedures, taking the kind of tablets they did not take during the first 8-week treatment period.

We will compare the frequency of urination, sleep, mood as adjusted for the tendency to make positive or negative judgments and daytime attention level to find if any of these differ between the two treatment periods, and to explain differences between any differences that may be found.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menopausal women, age 45 to 65 years old.
2. No menses for at least 6 months before the study start.
3. Have at least 14 episodes of nocturia per week.
4. Have at least 4 hot flashes daily.
5. Overall good health, as evidenced by a letter from the primary care provider.
6. Agree not to use exogenous hormones including soy isoflavones or soybean-based shakes, or nutritional supplements that potentially reduce hot flashes.
7. Have discontinued all hormone treatments, systemic, topical, or vaginal, at least 60 days before admission and throughout participation in the study.

Exclusion Criteria:

1. Use of anti-cholinergic, hypnotic or sedating drugs
2. Presence of urinary retention, gastric retention, chronic severe constipation,or narrow-angled glaucoma.
3. A urinary tract infection within a month of study start.
4. Undiagnosed abnormal vaginal bleeding.
5. Benign or malignant liver disease.
6. History or presence of chronic alcoholism or medication addiction within the past 5 yrs.
7. An acute systemic infection within seven days before the study start.
8. Concurrent participation in another clinical trial and/or receiving an experimental medication/device in the last 30 days before admission to the study.
9. History of shift work within the past 6 months.

   -

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-04; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quentin R Regestein, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Roehrs T, Merlotti L, Petrucelli N, Stepanski E, Roth T. Experimental sleep fragmentation. Sleep. 1994 Aug;17(5):438-43. doi: 10.1093/sleep/17.5.438. PMID 7991955
- [Background] Shaver JL, Paulsen VM. Sleep, psychological distress, and somatic symptoms in perimenopausal women. Fam Pract Res J. 1993 Dec;13(4):373-84. PMID 8285088
- [Background] Ancoli-Israel S, Cole R, Alessi C, Chambers M, Moorcroft W, Pollak CP. The role of actigraphy in the study of sleep and circadian rhythms. Sleep. 2003 May 1;26(3):342-92. doi: 10.1093/sleep/26.3.342. PMID 12749557
- [Background] Brooks JO 3rd, Friedman L, Bliwise DL, Yesavage JA. Use of the wrist actigraph to study insomnia in older adults. Sleep. 1993 Feb;16(2):151-5. doi: 10.1093/sleep/16.2.151. PMID 8446835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women 45 to 65 years old were mailed post-cards with the study telephone number and e-mail address. Subjects were assessed for eligibility. The PI determined eligibility based on the study criteria. Eligible subjects were informed about the study requirements, risks and benefits, and then required to read and sign a consent form.
Pre-assignment Details: Placebo responders were excluded after one week.
Period: Overall Study
Arm/Group | Tolterodine | Placebo
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolterodine | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (5.2) | 53 (5.2) | 52 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Nocturnal Urinary Frequency, Recorded on an Event/Symptom Chart;
Description: Subjects note: 1. Number of nocturnal and diurnal voids; 2) level of urgency for 7 days, graded 1 to 4, beginning after the first void on the Friday morning of week 7 and week 13 of their participation; 3) Number of incontinence episodes; 4) Relationship of incontinence to urge or stress (4 grade scale); 4) Whether she used any pads.
Time Frame: 2 months
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Urgency
Description: Level of urgency for 7 days, graded 1 to 4,
Time Frame: Beginning after the first void on the Friday morning of week 7 and week 13 of their participation;
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Incontinence Episodes;
Description: Number
Time Frame: Duration of Study
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Relationship of Incontinence to Urge or Stress
Description: 4-grade scale
Time Frame: Duration of study
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Psychological Self-reports, Scores on Anxiety and Depression Rating Scales;
Description: State and Trait scores on Spielberger State-Trait Anxiety Inventory; The score measured by the Zung Self-Rating Depression Inventory.
Time Frame: 2 weeks
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Quality of Life, Scores on the Women's Health Questionnaire.
Description: Self-reported vasomotor symptoms, other somatic symptoms, anxiety, depression, sleep and cognitive symptoms (memory, concentration and clumsiness problems), measured as category scores. Subjective sleep onset and total sleep times measured as 7-day averaged minutes.
Time Frame: 2 weeks
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Sleep Quality
Time Frame: 2 months
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Cognitive Function
Description: Motor speed (number of finger taps in 30 seconds); Continuous Performance (mean response time elicited by appearance of target alphabet letter presented in a series of letters on a monitor screen for 1 minute); Color-Word Stroop Test (response times to stimuli with congruent word and color)
Time Frame: Two 20-minute sessions during 2 months
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Hyperarousal
Description: Score on 26-item self-report Hyperarousal Scale that indicates proportion of attention allocated to visceral-somatic information vs. external sensory data.
Time Frame: At baseline and 8 weeks later
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Whether She Used Any Pads.
Description: Yes/No
Time Frame: Duration of Study
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Pads Used
Description: Pads used
Time Frame: Duration of Study
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Sleep / Wake Pattern
Description: Wrist actigraphy measures of total daytime and nighttime activity scored by standardized Actiwatch measures of sleep and sake.
Time Frame: Two weeks
Population: No data collected or analyzed for the outcome measures.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: Only serious adverse effects were collected
Arm/Group | Tolterodine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/9
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolterodine (N=10) | Placebo (N=9)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Dropout patient explained she had to go to hospital because of pneumonia. However, tt remained unclear whether she in fact had pneumonia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No